CLINICAL TRIAL: NCT07383298
Title: Observational Study on Dose Optimization of Olverembatinib in Patients With Chronic Myeloid Leukemia in Chronic or Accelerated Phase
Status: Enrolling by invitation | Type: Observational
Sponsor: Qian Jiang (Other)
Responsible Party: Sponsor-Investigator, Qian Jiang, Professor, Deputy Chair, Department of Hematology, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: 2025PHB563-001
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; Olverembatinib; Dose Optimization
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — olverembatinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Olverembatinib 20mg — Olverembatinib dose reduction to 20 mg every other day after achieving CCyR or BCR::ABL1 (IS) ≤1% in patients with chronic myeloid leukemia in chronic phase or accelerated phase.

SUMMARY:
This study is a multicenter observational study aimed to investigate the efficacy and safety of olverembatinib dose reduction to 20 mg every other day (QOD) in patients with chronic myeloid leukemia (CML) in chronic phase or accelerated phase who have achieved complete cytogenetic response (CCyR) or BCR::ABL1 (IS) ≤1%. Approximately 100 cases are planned to be enrolled.Primary endpoint: Maintenance rate of CCyR or BCR::ABL1 (IS) ≤1% within 12 months.

Secondary endpoints: Cumulative major molecular response (MMR) rate, cumulative MR4 rate, cumulative MR4.5 rate, MMR loss-free survival rate, MR4 loss-free survival rate, treatment failure-free survival rate, progression-free survival rate, overall survival rate, and safety.

Data analysis will be performed using SAS version 9.4 and R version 4.1.2. The loss-free survival rates will be calculated using the Log-rank and Kaplan-Meier methods. The cumulative response achievement rates will be calculated using the Fine-Gray method. Multivariate analysis will employ COX regression to identify relevant risk factors significantly affecting time-to-event variables, with hazard ratios (HR) and confidence intervals calculated. All adverse events occurring in subjects during the clinical trial period will be observed, including abnormal clinical symptoms, vital signs, and laboratory findings, with documentation of their clinical manifestation characteristics, severity, onset time, duration, management, and prognosis, and assessment of their relationship with the study drug. The plan is to enroll 100 cases within 12-24 months, with at least 12 months of observation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Diagnosed with chronic myeloid leukemia in the chronic phase, currently receiving olverembatinib 30 mg or 40 mg every other day (QOD). The patient must have achieved and maintained at least two consecutive confirmations of complete cytogenetic response (CCyR) or BCR::ABL1 (IS) ≤ 1% prior to enrollment and has decided to switch to olverembatinib 20 mg QOD.
3. Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score of 0 to 2.
4. Signed informed consent must be obtained prior to any study-specific procedures. If the patient is unable to sign due to their medical condition, informed consent may be provided by the legal guardian or an immediate family member.
5. Subjects must be willing and able to comply with all study procedures and the follow-up schedule.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

* Female patients with a positive serum β-HCG test, or who are pregnant, breastfeeding, or planning to become pregnant during the study period;

  * Uncontrolled infection at the time of enrollment; or severe complications requiring mechanical ventilatory support or presenting with hemodynamic instability; ③ Inability or unwillingness to provide signed informed consent; ④ Any condition or disease that, in the judgment of the investigator, may compromise subject safety or interfere with the evaluation of the efficacy or safety of the investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic myeloid leukemia in chronic phase or accelerated phase received olverembatinib
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
12-month CCyR or BCR::ABL1 ≤1% rate | 12 month
  12-month CCyR or BCR::ABL1 ≤1% rate

SECONDARY OUTCOMES:
Cumulative MMR rate | 24 months
  Cumulative MMR rate
Cumulative MR4 rate | 24 months
  Cumulative MR4 rate
Cardiovascular and cerebrovascular events | 24 month
  Cardiovascular and cerebrovascular events
Quality of life by EORTC QLQ-C30 | 24 months
  Quality of life by EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Qian Jiang, Dr., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available for sharing.
Supporting Information: Study Protocol
Time Frame: Upon article publication
Access Criteria: Access to the individual participant data (IPD) and supporting information will be granted to:
  Qualified researchers, including academic and clinical investigators Individuals or teams affiliated with recognized research, healthcare, or regulatory institutions Requestors who provide a valid, scientifically sound research proposal aligned with ethical guidelines and approved by an independent review committee (e.g., an institutional review board or ethics committee) Requestors who commit to using the data only for the approved research purpose and agree to applicable terms of data use